CLINICAL TRIAL: NCT04002791
Title: Randomized COmparison of Isolated Radial Artery ComPrEssioN Versus Radial and Ipsilateral Ulnar Artery Compression in Achieving Patent Hemostasis: OPEN-Radial Trial
Brief Title: Patent Hemostasis With Vasoband Versus TR Band
Acronym: OPEN-Radial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Total Cardiovascular Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A98
Record Dates: First submitted 2019-05-10; First posted 2019-07-01 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Radial Artery Injury at Wrist and Hand Level

STUDY DESIGN:
Intervention Model Description: Randomized comparison of patent hemostasis achievement with single bladder radial artery compression device with a dual-bladder ulnar compression capable radial artery compression device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1: TR Band Arm (Placebo Comparator): Patients will receive hemostatic compression using the current standard of care TR band (Terumo Corporation, Japan). The band will be applied according to the instructions for use, with optimal pressure applied using "Patent hemostasis protocol" to achieve full hemostasis.
  Interventions: Device: VasoBand
- Group 2: Vaso-band Arm (Active Comparator): Patients will receive Vaso-band (VasoInnovations, Inc, USA), applied with ulnar balloon inflated with 15 ml of air, and the radial balloon inflated after the sheath is removed, to apply optimal pressure for obtaining full hemostasis. Ulnar balloon will be deflated after 60 minutes of radial artery hemostatic compression.
  Interventions: Device: VasoBand

INTERVENTIONS:
Device: VasoBand — Dual-bladder radial artery hemostatic compression device capable of ipsilateral ulnar artery compression

SUMMARY:
In patients referred for cardiac catheterization to be performed using transradial access, a randomized comparison will be performed with the primary endpoint of patency of radial artery at the time of application of hemostatic compression band. The single radial only TR-Band (Terumo, Japan) will be compared to the dual balloon Vasoband (Vasoinnovations, USA) capable of ipsilateral ulnar artery compression.

DETAILED DESCRIPTION:
Introduction:

TRA is increasing in utilization across the world due to its established benefits of reduction in access site complications, cost, and increase in patient comfort (1). The most common structural consequence of TRA is radial artery occlusion (RAO). It occurs in 2-10% of patients undergoing TRA (2). Several pharmacologic as well as non-pharmacologic practices have been associated with RAO. Maintaining a hardware profile smaller than the inner diameter of radial artery has been associated with better radial artery patency rates after the procedure (3). Use of unfractionated heparin and other parenteral anticoagulants administered during the procedure has also been associated with reduction in RAO, with a dose-dependent effect with better reduction with higher doses of heparin (4,5).

One of the most effective intervention for reduction of RAO is avoidance of flow cessation in radial artery during hemostatic compression (6). This technique, called "patent hemostasis", has been shown to unequivocally and sizably reduce the incidence of RAO. In patients with small diameter radial arteries as well as low blood pressures, the ability to achieve and maintain patent hemostasis has been observed to be lower than those otherwise. In view of the co-dominant nature of forearm arterial circulation, the radial and ulnar arteries are interdependent and compression of ipsilateral ulnar artery has been shown to increase flow as well as peak flow velocity in the radial artery (7). Ipsilateral ulnar artery compression during hemostatic compression of a punctured radial artery, has been shown to sizably and significantly reduce the incidence of RAO compared to patent hemostasis (8). Randomized and observational datasets utilizing this technique published so far have been using two devices to achieve radial and ulnar compression, with difficult ergonomics leading to frequent dislodgment of ulnar compression during the radial artery hemostatic process.

The investigators intend to study the comparative efficacy of the first dedicated dual compression device in achieving patent hemostasis compared to the current popular radial artery compression device.

Patients and Methods:

Patients referred for diagnostic cardiac catheterization using TRA will be screened. Those providing written informed consent, will be enrolled in the study. A transradial cardiac catheterization will be performed using the standard technique as described below.

Catheterization Technique:

After sterile preparation as well as local anesthetic infiltration, 5 French hydrophilic introducer sheath will be introduced in the radial artery using standard puncture technique (9). Once the introducer is in the radial artery lumen, 200 µg of nitroglycerin, 2.5 mg of verapamil and 5000 IU of unfractionated heparin will be administered intra-arterially. 5 French or lower profile hardware will be used as per operator discretion to complete the procedure.

Once the procedure is completed, the patient will be randomized to:

Group 1, which will include patients receiving hemostatic compression using the current standard of care TR band (Terumo Corporation, Japan). The band will be applied according to the instructions for use, with optimal pressure applied to achieve full hemostasis.

Group 2, will consist of patients who will receive Vaso-band (VasoInnovations, Inc, USA), applied according to instructions for use, with ulnar balloon inflated for the first 60 minutes of radial artery hemostatic compression, with the radial balloon inflated to obtain full hemostasis, after the sheath is removed.

Primary Study End-point: Radial artery patency at 0-15 minutes after application of radial artery hemostatic compression.

Monitoring of Patency:

The radial artery patency will be monitored immediately after application of the band using reverse Barbeau test in both groups, and patency will be re-evaluated at 15 minutes after band application, 30 minutes after band application, 60 minutes after band application, as well as upon removal of the band at 120 minutes.

If longer duration of application of pressure with the band is necessary in either group to achieve hemostasis, the bands will be applied for longer duration and the adequacy of hemostasis will be evaluated every 15 minutes after 120-minute duration and the band removed once adequately adequate hemostasis has been achieved.

Radial patency will be assessed at 60 minutes after the band is removed.

Baseline demographic as well as procedural data, pharmacologic data, as well as elaborately data will be collected on every patient.

Statistical Analysis Plan:

Categorical variables will be expressed as proportions, and differences between the two groups will be assessed using chi-square test, or Pearson test as deemed appropriate. Numeric variables will be assessed for normality of the distribution, and will be expressed as mean and standard deviation for normally distributed variables, and median as well as interquartile range for those without normal distribution. Parametric tests will be used to compare differences between the two groups for normally distributed numeric variables, and nonparametric tests will be used in those variables with a non-normal distribution. Multivariable analysis if necessary, will be performed using forward selection binary logistic regression for categorical dependent variable and linear regression for numeric variables. Received operative characteristic derived c-statistic will be used to assess the stability of the model.

Sample Size Calculation:

Based on the available literature, using the current standard of care TR band, patent hemostasis defined as patency of radial artery during hemostatic compression at 15 minutes into compression is achievable in 75% of patients undergoing TRA. The only published randomized trial using prophylactic ipsilateral ulnar artery compression during radial artery hemostatic compression has shown 96% achievement of patent hemostasis at 15 minutes after onset of compression. Using this using these data, using a chi-square model, a sample size of 250 to 300 patients equally divided between two groups, is necessary to achieve a 90% power with an alpha editor of 0.05. Expecting a 10% crossover rate will be accommodated a sample size of 200 patients will be needed. After randomizing 200 patients, an interim analysis will be performed. If event rates are low, the sample-size will be increased to 350 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for cardiac catheterization undergoing transradial access

Exclusion Criteria:

* Previous ipsilateral radial artery cannulation, oral systemic anticoagulation therapy, thrombolytic therapy in the previous 7 days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2019-03-16 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tejas M Patel, MD, Principal Investigator — Apex Heart Institute, Ahmedabad, India
Locations (1):
- Apex Heart Institute, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be deidentified and will not be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: TR Band Arm | Group 2: Vaso-band Arm
Started | 127 | 126
Completed | 127 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: TR Band Arm | Group 2: Vaso-band Arm | Total
Number analyzed (Participants) | 127 | 126 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 59 (11) | 58 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 33 | 72
  Male | 88 | 93 | 181
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  INDIAN | 127 | 126 | 253
Hypertension [Count of Participants; unit: Participants] | 80 | 79 | 159
Diabetes [Count of Participants; unit: Participants] | 49 | 46 | 95
Previous PCI [Count of Participants; unit: Participants] | 12 | 12 | 24
Previous CABG [Count of Participants; unit: Participants] | 1 | 4 | 5
Height [Median (Inter-Quartile Range); unit: Centimeter] | 165 [160 to 170] | 165 [159 to 170] | 165 [160 to 170]
Weight [Median (Inter-Quartile Range); unit: Kilograms] | 72 [65 to 80] | 71 [65 to 80] | 71 [65 to 80]
Hemoglobin [Median (Inter-Quartile Range); unit: Gram/Dl] | 13.5 [12 to 14.8] | 13.2 [12.2 to 14.2] | 13.3 [12.2 to 14.5]
Platelets [Median (Inter-Quartile Range); unit: Cells x1000/ml] | 270 [209.5 to 322.5] | 250.5 [214.8 to 310.2] | 261 [214 to 318.5]
Serum Creatinine [Median (Inter-Quartile Range); unit: mg/dl] | 0.91 [0.76 to 1] | 0.91 [0.75 to 1.1] | 0.91 [0.75 to 1.05]
Wrist Circumference [Median (Inter-Quartile Range); unit: cm] | 21 [20 to 23] | 20 [19 to 23] | 20 [19 to 23]
Barbeau Test Pattern A [Count of Participants; unit: Participants] — Barbeau Test is performed by placing a plethysmographic sensor on the index finger after which the radial artery is compressed to the point of occlusion, and the plethysmographic waveform is analyzed, categorized into 4 categories.
  Pattern A is when the waveform shows no change from its baseline. Pattern B is when the waveform shows a decrease in amplitude from its baseline. Pattern C is when the waveform disappears but returns in < 2 minutes. Pattern D is when the waveform disappears and fails to return in < 2 minutes.
  Participants | 70 | 75 | 145
Barbeau Test Pattern B [Count of Participants; unit: Participants] — Barbeau Test is performed by placing a plethysmographic sensor on the index finger after which the radial artery is compressed to the point of occlusion, and the plethysmographic waveform is analyzed, categorized into 4 categories.
  Pattern A is when the waveform shows no change from its baseline. Pattern B is when the waveform shows a decrease in amplitude from its baseline. Pattern C is when the waveform disappears but returns in < 2 minutes. Pattern D is when the waveform disappears and fails to return in < 2 minutes.
  Participants | 53 | 46 | 99
Barbeau Test Pattern C [Count of Participants; unit: Participants] — Barbeau Test is performed by placing a plethysmographic sensor on the index finger after which the radial artery is compressed to the point of occlusion, and the plethysmographic waveform is analyzed, categorized into 4 categories.
  Pattern A is when the waveform shows no change from its baseline. Pattern B is when the waveform shows a decrease in amplitude from its baseline. Pattern C is when the waveform disappears but returns in < 2 minutes. Pattern D is when the waveform disappears and fails to return in < 2 minutes.
  Participants | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved Patent Hemostasis
Description: Patent hemostasis achievement at 0-15 minutes after onset of radial artery hemostatic compression
Time Frame: 0-15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: TR Band Arm | Group 2: Vaso-band Arm
Number analyzed (Participants) | 127 | 126
Participants | 94 | 122

2. Secondary Outcome: Number of Participants With Radial Artery Occlusion One Hour After Removal of Hemostatic Compression
Description: Absence of Patency of radial artery at 1-hour after removal of hemostatic compression
Time Frame: 0-60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: TR Band Arm | Group 2: Vaso-band Arm
Number analyzed (Participants) | 127 | 126
Participants | 13 | 2

ADVERSE EVENTS:
Time Frame: The event of Forearm Hematoma was assessed in the time period of the procedure, from the point of obtaining arterial access to the point of discharge from the catheterization laboratory, up to 4 hours or similar The event of Rebound Bleeding was assessed in the time period after removal of hemostatic compression band up to 1 hour or similar which is typically 4 hours or similar from the time of arterial puncture.
Description: Forearm Hematoma is a new swelling in the forearm as a result of bleeding Rebound Bleeding is bleeding restarting at the access site after hemostasis was achieved
Arm/Group | Group 1: TR Band Arm | Group 2: Vaso-band Arm
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/126
Serious Adverse Events (participants affected / at risk) | 16/127 | 2/126
Other Adverse Events (participants affected / at risk) | 0/127 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: TR Band Arm (N=127) | Group 2: Vaso-band Arm (N=126)
Forearm Hematoma (Surgical and medical procedures) | 6 (6) | 0 (0)
Rebound Bleeding (Surgical and medical procedures) | 10 (10) | 2 (2)

LIMITATIONS AND CAVEATS:
Single-center, single-country study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04002791/Prot_SAP_002.pdf